CLINICAL TRIAL: NCT00658502
Title: Ocular Response Analyzer Assessment of Intraocular Pressure and Corneal Biomechanical Properties in Myopic and Anisometropic Patients Under Atropine Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shu-Wen Chang/Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: FEMH97006
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-03

CONDITIONS: Myopia; Anisometropia
MeSH Terms: conditions — Myopia; Anisometropia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Our study has three parts has three parts, and the main aim of the study is to find out if corneal hysteresis was associated with myopia or even a predictor of myopia poor control predictor:

* Part 1 of our study: patients with anisomeropia whose spherical equivalent refraction as measured by cycloplegic autorefraction between the two eyes differ greater than 1.5 D.
* Part 2 of our study: Minus spherical equivalent refraction as measured by cycloplegic autorefraction.
* Part 3 of our study: patients with minus spherical equivalent refraction as measured by cycloplegic autorefraction who are under regular atropine for the treatment of myopia;patients who are prescribed with atropine treatment are in need of myopia control instead of for research interest

ELIGIBILITY:
Inclusion Criteria:

1. Normal ocular health other than myopia or anisometropia
2. In good general health with no history of prematurity or cardiac or significant respiratory diseases
3. No allergy to atropine, tropicamide, proparacaine, and benzalkonium chloride
4. No previous or current use of contact lenses, bifocals, progressive addition lenses
5. No amblyopia or manifest strabismus, including intermittent tropia

Exclusion Criteria:

1. presence of keratoconus or other corneal disease
2. previous eye drops usage except Atropine
3. major ocular surgery history (including refractive surgery, scleral buckle, glaucoma filtering, cornea transplant, cataract and vitreoretinal surgery)
4. presence of other ocular conditions such as glaucoma, uveitis, or other ocular inflammatory or vitreoretinal diseases.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: age under 25 year old with or without myopia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
axial length, corneal hysteresis | 3 month

SECONDARY OUTCOMES:
Refractive error, visual acuity, , intraocular pressure, , and corneal thickness | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan